CLINICAL TRIAL: NCT05737342
Title: Effect of ANKASCIN 568-P Products on Decreasing HbA1c and Regulating Blood Glucose- A Double-blind, Placebo-controlled Clinical Research
Brief Title: Effect of ANKASCIN 568-P Products on Decreasing HbA1c and Regulating Blood Glucose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22 ANKASCIN 568-P
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: High Blood Sugar; Metabolic Syndrome
MeSH Terms: conditions — Hyperglycemia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This experiment adopts a block random assignment design, and the system assignment table (Block randomization, block size = 6) randomly generated by the program is given serial numbers and assigned to groups. The probability of assignment to each group is 1/2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANKASCIN 568-P Red yeast rice capsules (Experimental): ANKASCIN 568-P is a fermented product from the red yeast rice fungus <Monascus purpureus NTU 568>. It does not contain Monacolin K, an ingredient that may harm the human body, and is rich in new active ingredients. Take 2 red yeast rice capsules (each containing 440mg ANKASCIN 568-P) every day, and the control group takes 2 placebo capsules (containing equal weight maltodextrin) every day, respectively, at the 0th, 4th , , 12, 24, Collect blood samples for biochemical analysis and record the general body position measurement, blood pressure, blood lipid, blood sugar and other related changes of the subjects, and monitor the liver, kidney, and thyroid functions.
  Interventions: Dietary Supplement: ANKASCIN 568-P Red yeast rice capsules
- Placebo Capsules (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: ANKASCIN 568-P Red yeast rice capsules — Product ingredients: ANKASCIN 568-P red yeast rice product 440 mg,microcrystalline ,cellulose,Maltodextrin; capsule shell composition: HPMC (hydroxypropyl methylcellulose), purified water, titanium dioxide, gellan gum.
  Arms: ANKASCIN 568-P Red yeast rice capsules
Dietary Supplement: Placebo Capsules — Maltodextrin was used as a placebo
  Arms: Placebo Capsules

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-controlled trial (24 weeks in total), divided into three periods (screening, treatment, and discontinuation follow-up)

DETAILED DESCRIPTION:
This trial is a randomized double-blind human trial, mainly to investigate the effect of long-term consumption of red yeast rice products on reducing glycated hemoglobin (HbA1c) and regulating blood sugar. It is expected to recruit 80 subjects for a period of 24 weeks. The test group takes 2 capsules of red yeast rice per day (Each capsule contains 440mg ANKASCIN 568-P), the control group took placebo capsules daily, blood samples were collected for biochemical analysis at 0, 4, 12, and 24 weeks, and the general body position measurement, blood pressure, Blood lipids, blood sugar and other related changes, and monitor liver, kidney, thyroid function.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women over 20 years old (women of childbearing age are not allowed to become pregnant or breastfeed during the study) adults who are sane and able to communicate.
2. 18≦BMI≦35.
3. Blood routine examination (CBC; Complete blood count): the mean corpuscular volume MCV should not be less than 70 fL.
4. Blood glucose level measurement meets any of the following conditions:

(1) The fasting blood sugar is between 100∼125 mg/dL, and the doctor judges that there is no need to use hypoglycemic drugs for the time being.

(2) Or the glycosylated hemoglobin is between 5.7∼6.4%, and the doctor judges that the use of hypoglycemic drugs is not needed for the time being.

(3) Diabetic patients who have no willingness to take medicine and have not taken hypoglycemic drugs in the past month.

5. Those without other serious diseases (cancer, heart failure, myocardial infarction, liver cirrhosis, moderate to severe liver and kidney dysfunction, stroke, etc.).

6. Hypoglycemic drugs are not allowed to be used during the trial. If the condition changes and the use of hypoglycemic drugs is required, the trial must be withdrawn.

7. During the test period, the daily routine and eating habits should be maintained without deliberately changing them.

Exclusion Criteria:

1. Blood pressure: systolic blood pressure ≧ 200 mmHg or diastolic blood pressure ≧ 140 mmHg.
2. Moderate or severe liver and kidney dysfunction (generally refers to serum aminopyruvate converting enzyme (SGPT) and serum glutamate phenylacetate transaminase (SGOT) are more than 3 times higher than the upper limit of normal value or have been diagnosed Liver cirrhosis, or glomerular filtration rate eGFR≦30 ml/min/1.73m2).
3. Pregnant or lactating women.
4. Diabetic patients taking hypoglycemic drugs or insulin injections.
5. Those who take traditional Chinese medicine mainly red yeast rice.
6. Have undergone surgery within one month.
7. Combined with serious diseases such as heart, liver, kidney and hematopoietic system, mentally ill patients who do not meet the inclusion criteria, who do not eat the test samples according to the regulations, so that the efficacy cannot be judged or the incomplete data affect the judgment of efficacy or safety.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Improve glycated hemoglobin (HbA1c) value | 24 weeks
  After 24 weeks of taking red yeast rice capsules or placebo gel, whether there is a statistical difference between the test group and the placebo group in terms of improving the HbA1c value of glycosylated hemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: WEN-HUI FANG, Ph. D., Principal Investigator — Chief of Family medicine department
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei city,, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hsu LC, Hsu YW, Hong CC, Pan TM. Safety and mutagenicity evaluation of red mold dioscorea fermented from Monascus purpureus NTU 568. Food Chem Toxicol. 2014 May;67:161-8. doi: 10.1016/j.fct.2014.02.033. Epub 2014 Feb 28. PMID 24582683
- [Result] Shi YC, Pan TM. Anti-diabetic effects of Monascus purpureus NTU 568 fermented products on streptozotocin-induced diabetic rats. J Agric Food Chem. 2010 Jul 14;58(13):7634-40. doi: 10.1021/jf101194f. PMID 20557124
- [Result] Shi YC, Pan TM. Antioxidant and pancreas-protective effect of red mold fermented products on streptozotocin-induced diabetic rats. J Sci Food Agric. 2010 Nov;90(14):2519-25. doi: 10.1002/jsfa.4115. PMID 20737515
- [Result] Shi YC, Liao JW, Pan TM. Antihypertriglyceridemia and anti-inflammatory activities of monascus-fermented dioscorea in streptozotocin-induced diabetic rats. Exp Diabetes Res. 2011;2011:710635. doi: 10.1155/2011/710635. Epub 2011 May 11. PMID 21716679
- [Result] Lee BH, Hsu WH, Huang T, Chang YY, Hsu YW, Pan TM. Monascin improves diabetes and dyslipidemia by regulating PPARgamma and inhibiting lipogenesis in fructose-rich diet-induced C57BL/6 mice. Food Funct. 2013 Jun;4(6):950-9. doi: 10.1039/c3fo60062a. Epub 2013 May 14. PMID 23673903
- [Result] Chen CL, Pan TM. Effects of red mold dioscorea with pioglitazone, a potentially functional food, in the treatment of diabetes. J Food Drug Anal. 2015 Dec;23(4):719-728. doi: 10.1016/j.jfda.2015.04.013. Epub 2015 Jul 21. PMID 28911488
- [Result] Slim R, Ben Salem C, Zamy M, Biour M. Pioglitazone-induced acute rhabdomyolysis. Diabetes Care. 2009 Jul;32(7):e84. doi: 10.2337/dc09-0593. No abstract available. PMID 19564463
- [Result] Wang YR, Liu SF, Shen YC, Chen CL, Huang CN, Pan TM, Wang CK. A randomized, double-blind clinical study to determine the effect of ANKASCIN 568 plus on blood glucose regulation. J Food Drug Anal. 2017 Apr;25(2):409-416. doi: 10.1016/j.jfda.2016.06.011. Epub 2016 Jul 30. PMID 28911684
- [Result] Liu SF, Wang YR, Shen YC, Chen CL, Huang CN, Pan TM, Wang CK. A randomized, double-blind clinical study of the effects of Ankascin 568 plus on blood lipid regulation. J Food Drug Anal. 2018 Jan;26(1):393-400. doi: 10.1016/j.jfda.2017.04.006. Epub 2017 Jun 1. PMID 29389579